CLINICAL TRIAL: NCT05424536
Title: Cortical Bone Assessment Using Ultrasonic Guided Waves: Towards a Robust Clinical
Brief Title: Cortical Bone Assessment Using Ultrasonic Guided Waves: Towards a Robust Clinical Measurement
Acronym: BDATChile
Status: Completed | Type: Observational
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Pontificia Universidad Catolica de Valparaiso (Other); Centro Gerópolis UV, Valparaíso (Unknown); Centro de Salud Familiar Marcelo Mena (Unknown); Hospital Dr. Gustavo Fricke, Valparaíso (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1201311
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2023-01

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bone measurement by DXA and ultrasound — Measurement will be performed at radius and at tibia (ultra-distal and distal). For all the sites plus femoral neck, one measurement will be performed by DXA to get reference values of thickness and BMDs. For the distal positions and additional measurement will be performed by an innovative ultrasound device that estimates cortical thickness and porosity.

SUMMARY:
Osteoporosis is a skeletal disease leading to bone fragility and increasing the risk of fractures and still remains a major public health problem worldwide. Therefore it is crucial to prevent severe fractures responsible for excess of mortality and considerable morbidity. Patient at risk of fractures are currently identified as having osteoporosis using Dual-energy X-ray Absorptiometry (DXA), assessing the areal or projected Bone Mineral Density (aBMD g.cm-2). In Chile, the hip fracture occurrence is very similar to the international incidence. Due to the demographic and epidemiological transition, the number of hip fracture for patient older than 50 year, is expected to severely increase from about 6.500 (2007) to 30.000 (2050) without adequate preventive and / or therapeutic measures.

Even if DXA remains the current gold standard, it is limited by the difficulty to set a threshold in the BMD distribution for osteoporosis diagnosis. Moreover, some medical conditions (chronic kidney disease, diabetes) or drugs (glucocorticoids) are associated with an increase of fracture risk without a BMD decrease. Quantitative ultrasound (QUS) have the advantages of portability, low cost, absence of radiation and need for a radiographic technologist or designated room, and are sensitive to both elasticity and geometry of the medium explored by the waves. Among QUS techniques, axial transmission (AT) is a technique for which transducers are aligned along the bone axis. Measured ultrasonic guided waves, associated with an appropriate waveguide model have the potential to yield estimates of material and/or geometrical cortical properties. In vivo combined estimation of both cortical thickness and porosity has been proposed using bidirectional axial transmission (BDAT). BDAT measurement has been recently validated on ex vivo specimen (radius and tibia) and has been tested in a pilot clinical study, in which cortical porosity measured at the one-third distal radius has been found as discriminant of low trauma fractures as DXA. Cortical porosity is increasingly recognized as a major contributor to bone fragility.

The hypothesis underlying this project are that (1) it is possible to obtain robust and accurate estimates of cortical thickness and porosity using an improved BDAT device and (2) these estimates are of clinical interest in the context of osteoporosis in elderly. Moreover, novel parameters obtained from automatic classification tools will be tested.

DETAILED DESCRIPTION:
The purpose of this investigation is to determine if there are differences in the quantities of cortical bone (thickness and porosity) as well as the new parameters measured by BDAT at both forearm and leg, between patients with recent non traumatic fracture and controls.

Results will be compared to the current gold standard dual-energy X-ray absorptiometry (DXA) of the hip, spine and forearm, obtained from all subjects. The BDAT device with the improved interface will be tested in a clinical environment by clinical operators on:

* minimum sample size per group: 25 for cases and controls (female and male, over 50 years).
* Fractured patients will be obtained at the traumatology service of Fricke Hospital (Viña del Mar) which receives about 350 patients with hip fractures per year.
* Control will be obtained at the community health centers of Valparaiso in collaboration with the UV project Geropolis.

DXA measurement will be done at the imaging center of the Universidad Catolica de Valparaiso (PUCV, FONDEQUIP EQM160142). Additional DXA parameters concerning muscle and fat, will be taken into account.

ELIGIBILITY:
For both groups:

Inclusion Criteria:

* > 50 years old

Exclusion Criteria:

* History of fracture
* Corticoid treatment
* Renal disease
* Arthritis
* BMI < 15 and > 30
* Double femoral prosthesis

In case group/with fracture is added:

Inclusion criteria

* Recent femoral bone fragility fracture

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be:
  Women and men over 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Cortical parameter measurement obtained by BDAT (Ultrasound) | Inclusion time
  Cortical thickness (mm) at one-third distal radius and mid-tibia
Cortical parameter measurement obtained by BDAT (Ultrasound) | Inclusion time
  Cortical porosity (%) at one-third distal radius and mid-tibia
Ultrasonic velocities measurement obtained by BDAT (Ultrasound) | Inclusion time
  velocity (m.s-1) of the First Arriving Signal (VFAS) at one-third distal radius and mid-tibia
Ultrasonic velocities measurement obtained by BDAT (Ultrasound) | Inclusion time
  velocity (m.s-1) of the A0 guided mode (A0) at one-third distal radius and mid-tibia

SECONDARY OUTCOMES:
Quality measurement parameter obtained by BDAT (Ultrasound) | Inclusion time
  measurement at one-third distal radius and mid-tibia, normalized quality parameter (value ranging from 0 to 1).
femoral aBMD obtained by DXA | Inclusion time
  measurement of femoral areal Bone Mineral Density (aBMD g.cm-2).
Body composition measurements obtained by DXA | Inclusion time
  body composition: body fat, muscle and bone mass (kg).
10-year probability of fracture provided by FRAX algotithm | Inclusion time
  10-year probability of a major osteoporotic fracture, calculated with the femoral aBMD value.
10-year probability of fracture provided by FRAX algotithm | Inclusion time
  10-year probability of a major osteoporotic fracture, calculated without the femoral aBMD value.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Gabriel Minonzio, Ph.D, Principal Investigator — Universidad de Valparaiso; José Luis Dinamarca, M.D., Study Chair — Universidad de Valparaiso
Locations (1):
- Universidad de Valparaíso, Valparaíso, Chile

REFERENCES:
- See also: study using the same ultrasonic device — https://doi.org/10.1371/journal.pone.0277831
- See also: The FRAX® algorithms give the 10-year probability of fracture. — https://frax.shef.ac.uk/frax/